CLINICAL TRIAL: NCT04037397
Title: First Line Radiofrequency Ablation Versus Antiarrhythmic Drugs for Persistent Atrial Fibrillation Treatment
Brief Title: First Line Radiofrequency Ablation Versus Antiarrhythmic Drugs for Persistent Atrial Fibrillation Treatment (RAAFT-3)
Acronym: RAAFT-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Biosense Webster, Inc. (Industry); Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 829475
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
Keywords: Pulmonary Vein Isolation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Intervention Model Description: 120 patients will be randomized in a 2:1 fashion (80 in the RFCA arm; 40 in the AADs arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antiarrhythmic Medications (Active Comparator): Patients randomized to the antiarrhythmic drug group are administered medications approved for treatment of AF by the regulatory bodies of each participating country. The selection of antiarrhythmic drugs and dosages is left to the discretion of the investigator, and will follow the AHA/ACC/HRS general guidelines
  Interventions: Drug: Anti Arrhythmics
- Radio Frequency Catheter Ablation (Active Comparator): Patients randomized to radiofrequency catheter ablation will undergo isolation of the pulmonary veins with confirmation of entrance block into each vein. The CARTO TM(Biosense Webster, CA) system will be used to reconstruct the atrial geometry and assist for mapping and ablation. Ablation will be performed using approved ablation devices (Biosense Webster, CA).
  Interventions: Procedure: Pulmonary Vein Isolation performed by Radio Frequency Catheter Ablation

INTERVENTIONS:
Drug: Anti Arrhythmics — Propafenone or Flecanide or Sotalol or Dofetilide or Dronedarone or Amiodarone. The subject must first fail a Class 1C or III drug prior to starting Amiodarone
  Arms: Antiarrhythmic Medications
Procedure: Pulmonary Vein Isolation performed by Radio Frequency Catheter Ablation — Approved Biosense Webster Inc. catheter devices should be used to perform RFCA. Ablation will be done to achieve entrance block into all pulmonary veins
  Arms: Radio Frequency Catheter Ablation

SUMMARY:
The purpose of this study is to determine if catheter-based atrial fibrillation (AF) ablation is superior to treatment with antiarrhythmic drugs as a first-line therapy for symptomatic persistent AF.

DETAILED DESCRIPTION:
The burden of atrial fibrillation (AF) on Western countries healthcare systems is steadily increasing, with over 2 million Americans and 4 million Europeans affected by this condition. It is by far the most common sustained arrhythmia encountered in clinical practice, with a striking impact on morbidity and mortality. Achieving a definite cure is highly desirable, as this would have profound social and economic implication. In patients with drug-refractory paroxysmal AF, multiple clinical trials have established the superiority of catheter ablation over further antiarrhythmic drug (AAD) therapy for the long-term maintenance of sinus rhythm, to improve quality of life, and reduce hospitalizations. Recent randomized controlled trials have also demonstrated a beneficial role of catheter ablation as a first-line therapy in patients with paroxysmal AF, with significantly better arrhythmia control and improved quality of life compared to AAD therapy. Patients with symptomatic persistent AF represent a more challenging group to treat, given the overall lower success rate of catheter ablation procedures in this group of patients. Pharmacologic rhythm-control strategies are also less effective in persistent AF, with a substantially increased economic burden given the repeat admissions for electrical cardioversions and AAD initiation/titration. In patients with symptomatic persistent AF who have already failed AADs, catheter ablation has been shown superior to further AAD therapy for sinus rhythm restoration in a recent randomized controlled trial. However, the value of an upstream adoption of catheter ablation for the treatment of symptomatic persistent AF (i.e., before a trial with AADs) is unknown. The purpose of the third Radiofrequency Ablation vs Antiarrhythmic Drugs for Atrial Fibrillation Treatment (RAAFT-3) trial is to determine whether catheter ablation is superior to AAD as a first-line therapy in patients with persistent AF who had not been exposed to antiarrhythmic treatment.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients have a history of persistent AF with at least 2 episodes in the 9 months prior to enrollment. Persistent AF is defined according to 2014 AHA/ACC/HRS guidelines as continuous AF that is sustained for more than 7 days.Patients are enrolled if they are:

1. Older than 18.
2. Symptomatic with persistent AF.
3. Experienced at least one AF episode that was documented by surface ECG, 6 months before randomization.

Exclusion Criteria:

1. Documented LVEF <40%.
2. Documented left atrial diameter >/=6cm.
3. Moderate to severe LVH (LV wall thickness >1.5cm).
4. Documented severe valvular disease (aortic stenosis, mitral regurgitation, tricuspid regurgitation or presence of mechanical cardiac valves), active coronary artery disease (defined as the presence of >70% stenosis of coronary arteries or documentation of active myocardial ischemia), recent (within 6 months) CABG.
5. Untreated hypothyroidism or hyperthyroidism. Patients who are euthyroid on thyroid hormone replacement therapy are acceptable.
6. Contraindication for the use of all antiarrhythmic drugs including sotalol, dofetilide, amiodarone and 1C antiarrhythmic drugs (liver enzymes and serum creatinine that are outside the upper normal lab values, e.g. > 3 times ULN with 2 abnormal lab values). [Note: Participants will not be excluded if they are able to take any single or combination of drugs without contraindications]
7. Previous left heart ablation procedure, either by surgery or by percutaneous catheter, for atrial fibrillation.
8. Current enrollment in another investigational drug or device study.
9. Presence of any other condition that the investigator feels would be problematic or would restrict or limit the participation of the Patient for the entire study period.
10. Absolute contra-indication to the use of heparin and or oral anticoagulation.
11. Increase risk of bleeding, current peptic ulceration, proliferative diabetic retinopathy, history of severe systemic bleeding, or other history of bleeding diathesis or coagulopathy.
12. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD).
13. Documented intra-atrial thrombus, tumor, or another abnormality, which precludes left atrial catheter ablation.
14. Previous use of an antiarrhythmic drug, including amiodarone, propafenone, flecainide, sotalol, quinidine, dofetilide, dronedarone (see below for specifications: Antiarrhythmic Drug Group).
15. Women with a positive pregnancy test.
16. Evidence of active cardiac or systemic infection.
17. Medical condition limiting expected survival to less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of symptomatic Atrial Fibrillation | 18 Months
  Recurrence (post 90- day blanking period) of symptomatic or asymptomatic AF, atrial flutter, or atrial tachycardia lasting more than 30 seconds documented by the pre-defined ECG monitoring is the primary efficacy outcome. Any episodes occurring during the 90-day blanking period are not considered as recurrences

SECONDARY OUTCOMES:
Time to AF recurrence | 18 Months
  Time to first documented recurrence of AF, atrial flutter, and atrial tachycardia episodes
Repeat Episodes of AF | 18 Months
  Repeated episodes (≥2) of symptomatic or asymptomatic AF, atrial flutter, and atrial tachycardia episodes
AF/AT Burden | 18 Months
  Cumulative AF/AT burden (defined as percentage of time in AF/AT during follow-up)
CV Hospitalizations | 18 Months
  Hospitalization for cardiovascular and non-cardiovascular causes during follow-up
Quality of Life Questionnaire | 18 Months
  Quality of life at the 1-year follow-up by SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (5):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - Montefiore Medical Center, The Bronx, New York
  - MetroHealth, Cleveland, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Friberg J, Buch P, Scharling H, Gadsbphioll N, Jensen GB. Rising rates of hospital admissions for atrial fibrillation. Epidemiology. 2003 Nov;14(6):666-72. doi: 10.1097/01.ede.0000091649.26364.c0. PMID 14569181
- [Background] Bialy D, Lehmann H, Schumacher DN, Steinman RT, Meissner MD. Hospitalization for arrhythmias in the United States: importance of atrial fibrillation. J Am Coll Cardiol. 1992;19:41A
- [Background] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Background] Jais P, Cauchemez B, Macle L, Daoud E, Khairy P, Subbiah R, Hocini M, Extramiana F, Sacher F, Bordachar P, Klein G, Weerasooriya R, Clementy J, Haissaguerre M. Catheter ablation versus antiarrhythmic drugs for atrial fibrillation: the A4 study. Circulation. 2008 Dec 9;118(24):2498-505. doi: 10.1161/CIRCULATIONAHA.108.772582. Epub 2008 Nov 24. PMID 19029470
- [Background] Wazni OM, Marrouche NF, Martin DO, Verma A, Bhargava M, Saliba W, Bash D, Schweikert R, Brachmann J, Gunther J, Gutleben K, Pisano E, Potenza D, Fanelli R, Raviele A, Themistoclakis S, Rossillo A, Bonso A, Natale A. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of symptomatic atrial fibrillation: a randomized trial. JAMA. 2005 Jun 1;293(21):2634-40. doi: 10.1001/jama.293.21.2634. PMID 15928285
- [Background] Morillo CA, Verma A, Connolly SJ, Kuck KH, Nair GM, Champagne J, Sterns LD, Beresh H, Healey JS, Natale A; RAAFT-2 Investigators. Radiofrequency ablation vs antiarrhythmic drugs as first-line treatment of paroxysmal atrial fibrillation (RAAFT-2): a randomized trial. JAMA. 2014 Feb 19;311(7):692-700. doi: 10.1001/jama.2014.467. PMID 24549549
- [Background] Santangeli P, Di Biase L, Natale A. Ablation versus drugs: what is the best first-line therapy for paroxysmal atrial fibrillation? Antiarrhythmic drugs are outmoded and catheter ablation should be the first-line option for all patients with paroxysmal atrial fibrillation: pro. Circ Arrhythm Electrophysiol. 2014 Aug;7(4):739-46. doi: 10.1161/CIRCEP.113.000629. No abstract available. PMID 25140019
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Calkins H, Reynolds MR, Spector P, Sondhi M, Xu Y, Martin A, Williams CJ, Sledge I. Treatment of atrial fibrillation with antiarrhythmic drugs or radiofrequency ablation: two systematic literature reviews and meta-analyses. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):349-61. doi: 10.1161/CIRCEP.108.824789. Epub 2009 Jun 2. PMID 19808490
- [Background] Catherwood E, Fitzpatrick WD, Greenberg ML, Holzberger PT, Malenka DJ, Gerling BR, Birkmeyer JD. Cost-effectiveness of cardioversion and antiarrhythmic therapy in nonvalvular atrial fibrillation. Ann Intern Med. 1999 Apr 20;130(8):625-36. doi: 10.7326/0003-4819-130-8-199904200-00002. PMID 10215558
- [Background] Mont L, Bisbal F, Hernandez-Madrid A, Perez-Castellano N, Vinolas X, Arenal A, Arribas F, Fernandez-Lozano I, Bodegas A, Cobos A, Matia R, Perez-Villacastin J, Guerra JM, Avila P, Lopez-Gil M, Castro V, Arana JI, Brugada J; SARA investigators. Catheter ablation vs. antiarrhythmic drug treatment of persistent atrial fibrillation: a multicentre, randomized, controlled trial (SARA study). Eur Heart J. 2014 Feb;35(8):501-7. doi: 10.1093/eurheartj/eht457. Epub 2013 Oct 17. PMID 24135832
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883
- [Background] Macle L, Khairy P, Weerasooriya R, Novak P, Verma A, Willems S, Arentz T, Deisenhofer I, Veenhuyzen G, Scavee C, Jais P, Puererfellner H, Levesque S, Andrade JG, Rivard L, Guerra PG, Dubuc M, Thibault B, Talajic M, Roy D, Nattel S; ADVICE trial investigators. Adenosine-guided pulmonary vein isolation for the treatment of paroxysmal atrial fibrillation: an international, multicentre, randomised superiority trial. Lancet. 2015 Aug 15;386(9994):672-9. doi: 10.1016/S0140-6736(15)60026-5. Epub 2015 Jul 23. PMID 26211828
- [Background] Di Biase L, Santangeli P, Natale A. How to ablate long-standing persistent atrial fibrillation? Curr Opin Cardiol. 2013 Jan;28(1):26-35. doi: 10.1097/HCO.0b013e32835b59bb. PMID 23207492